CLINICAL TRIAL: NCT05329558
Title: Pilot Study: Local and Systemic Changes in Osteonecrosis of the Jawbone
Brief Title: Local and Systemic Changes in Osteonecrosis of the Jawbone
Acronym: SULVO
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Foessl, Ines, MSc, Investigator, Medical University of Graz
Other Study IDs: 30-196 ex 17/18
Record Dates: First submitted 2022-02-22; First posted 2022-04-15 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Osteonecrosis of the Jaw

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, plasma, serum, saliva, tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Controls
- Patients with ART without MRONJ
- Patients with oral ART with MRONJ
- Patients with intravenous ART with MRONJ

SUMMARY:
Osteonecrosis of the Jawbone (ONJ) is a serious complication of antiresorptive therapies (ARTs), for example with bisphosphonates or Denosumab. Especially long term treatment with intravenous antiresorptive agents causing lesions and, less frequent, also oral administration. This study aims at elucidating local and systemic changes in patients with ONJ.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* with/without ART
* with/without MRONJ

Exclusion Criteria:

* smoker (>10 cigarettes/day)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at the Department of Oral Surgery and Radiology, University Clinic for Oral and Maxillofacial Medicine, Graz, Austria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
target gene expression | through study completion, an average of 1 year
  differences in gene expression recorded by qPCR will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Acham, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria